CLINICAL TRIAL: NCT03677752
Title: Guided Participation to Positioning (GP_Posit) Intervention for Mothers of Preterm Infants in the Neonatal Intensive Care Unit for Maternal Sensitivity and Infant's Neurodevelopment: Randomized Pilot Trial
Brief Title: GP_Posit Intervention for Mothers of Preterm Infants for Maternal Sensitivity : Randomized Pilot Trial
Acronym: GP_Posit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Andréane Lavallée, Student, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2017-1540
Record Dates: First submitted 2018-08-01; First posted 2018-09-19 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Preterm Infant; Mothers; Parent-Child Relations; Child Development; Interaction, Mother-Infant
Keywords: Intervention; Maternal sensitivity; Neurodevelopment; Maternal stress; Maternal anxiety; Neonatal intensive care unit
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GP_Posit (Experimental): Participants allocated to this arm will receive the GP_Posit intervention.
  Interventions: Other: GP_Posit
- Control (No Intervention): Participants in the control arm will receive usual care.

INTERVENTIONS:
Other: GP_Posit — Mother-infant dyads allocated to this arm will receive the GP_Posit intervention. The intervention consists of a guided participation intervention to positioning. Mothers will meet with the intervention nurse twice a week for the two first weeks after birth and then one a week until the infant will reach 35 weeks of gestational age. During these encounters, mothers will learn how to interpret their infant's stress and stability cues and participate in his/her care and positioning while being guided by the intervention nurse.
  Other Names: Guided Participation intervention to positioning
  Arms: GP_Posit

SUMMARY:
The aim of this study is to evaluate the acceptability, feasibility and preliminary effects a GP_Posit intervention. GP_Posit is an intervention where mothers will learn how to participated in their preterm infant's care and positioning while being guided by a nurse. Preliminary effects will be estimated on maternal sensitivity, stress and anxiety as well as preterm infant's neurodevelopment.

ELIGIBILITY:
This study will recruit mother-infant dyads.

Inclusion Criteria for mothers:

* Understand, write and read French and/or English
* Are 18 years or older

Exclusion Criteria for mothers:

* Use drugs
* Have an instable mental health
* Give their newborn infant for adoption

Inclusion Criteria for preterm infants:

* Are born at 27 0/7 et 31 6/7 weeks of gestation
* Are hospitalized in the NICU for at least 4 weeks

Exclusion Criteria for preterm infants:

* Require surgery
* Have intraventricular haemorrhage (IVH) > grade 2
* Have congenital malformations

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
Compliance to the protocole | Through study completion, an average of 1 1/2 year.
  Compliance to the protocole to assess feasibility of the intervention GP_Posit and protocol. Research team will document aspects regarding % of recruitment, % of intervention delivered as planned, etc. through study completion. A threshold of 80% will be used to determine feasibility of the protocole elements.
Content analysis of acceptability questionnaires | When the infant reaches 36 weeks of gestational age (after the intervention that finished at 35 weeks of gestational age; before NICU discharge)
  Mothers' answers to acceptability questionnaires will be analyzed. This is a questionnaire built by the research team aimed at collecting narrative data regarding mother's acceptability of the intervention. Elements such as acceptability of the length of the intervention, frequency of encounters, etc. will be assessed.

SECONDARY OUTCOMES:
Mother-Infant interaction | When the infant reaches 36 weeks of gestational age (after the intervention; before NICU discharge)
  Filmed mother-infant feeding will be coded to assess mother-infant interaction between the mother and the infant and maternal sensitivity to her infant's cues using the Parent-Child Interaction - Feeding Scale. The score can vary from 0-76 and a higher score is better.
Parental beliefs about preterm infant and parental role | At entry in the study and when the infant reaches 36 weeks of gestational age (after the intervention that finished at 35 weeks of gestational age; before NICU discharge)
  Neonatal intensive care unit: parental beliefs scale (NICU:PBS). Scale range: Likert type scale (1 to 5) where a higher score indicates better beliefs. Scores can vary from 18 to 90.
General movement assessment (GMA) | When the infant reaches 36 weeks of gestational age (after the intervention that finished at 35 weeks of gestational age; before NICU discharge)
  General movements of infants will be analyzed in order to analyse preterm infant's neurodevelopment.
Electroencephalogram (EEG) | At entry in the study and when the infant reaches 36 weeks of gestational age (after the intervention that finished at 35 weeks of gestational age; before NICU discharge)
  Electrical activity in the preterm brain will be measured using 8 electrodes on the infant's heads and compared before and after the intervention + between groups. We will perform spectral analyses with multiscale entropy calculation and connectivity analyses in order to see synchrony using the phase slope index.

OTHER OUTCOMES:
Maternal Anxiety | At entry in the study and when the infant reaches 36 weeks of gestational age (after the intervention that finished at 35 weeks of gestational age; before NICU discharge)
  State-trait anxiety inventory (STAI). Likert type scale with scores ranging from 1 to 4. A higher score indicates a worst outcome (more anxiety). Total score can range from 20 to 80.
Maternal stress | At entry in the study and when the infant reaches 36 weeks of gestational age (after the intervention that finished at 35 weeks of gestational age; before NICU discharge)
  Parental stressor scale: NICU Scale range: Likert type scale (1 to 5) where a higher score indicates higher levels of stress. The three subscales will be reported independently. First subscale can vary from 0 to 25. Second subscale can vary from 0 to 70. Third subscale can vary from 0 to 35.

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Aita, PhD, Study Director — Université de Montréal
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lavallee A, Aita M, Bourbonnais A, De Clifford-Faugere G. Effectiveness of early interventions for parental sensitivity following preterm birth: a systematic review protocol. Syst Rev. 2017 Mar 23;6(1):62. doi: 10.1186/s13643-017-0459-x. PMID 28335806
- [Derived] Lavallee A, Aita M, Cote J, Bell L, Luu TM. A guided participation nursing intervention to theraupeutic positioning and care (GP_Posit) for mothers of preterm infants: protocol of a pilot randomized controlled trial. Pilot Feasibility Stud. 2020 May 26;6:77. doi: 10.1186/s40814-020-00601-5. eCollection 2020. PMID 32509322